CLINICAL TRIAL: NCT03121963
Title: Pain Management in Head and Neck Surgery Patients
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: This protocol was difficult to enroll into, and changes to personnel have made it difficult to main this study. Data collection was not completed and therefore, no data analysis was performed. The PI has made the decision to close this study.
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Erin Partington, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-170310004
Record Dates: First submitted 2017-04-17; First posted 2017-04-20 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Pain Management
MeSH Terms: conditions — Agnosia | interventions — Oxycodone; Acetaminophen; Gabapentin; Celecoxib; oxycodone-acetaminophen

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Group (Experimental): A combination regimen of oxycodone 5 mg Q6hr PRN, acetaminophen 650 mg Q6hr, celecoxib 400 mg BID post-operatively x 2 weeks, and gabapentin 400 mg loading dose, 300 mg TID to be started 1 week pre-operatively then continued post-operatively x 2 weeks.
  Interventions: Drug: Oxycodone; Drug: Acetaminophen; Drug: Gabapentin; Drug: Celecoxib
- Control Group (Active Comparator): A single medication regimen of hydrocodone-acetaminophen 7.5 mg Q6hr PRN post-operatively x 2 weeks.
  Interventions: Drug: Hydrocodone-Acetaminophen

INTERVENTIONS:
Drug: Oxycodone — oxycodone tablet
  Other Names: Oxycontin
  Arms: Treatment Group
Drug: Acetaminophen — acetaminophen tablet
  Other Names: Tylenol
  Arms: Treatment Group
Drug: Gabapentin — gabapentin tablet
  Other Names: Neurontin
  Arms: Treatment Group
Drug: Celecoxib — celecoxib tablet
  Other Names: Celebrex
  Arms: Treatment Group
Drug: Hydrocodone-Acetaminophen — hydrocodone 5 mg/acetaminophen 325 mg tablet
  Other Names: Norco
  Arms: Control Group

SUMMARY:
Our study aims to see if the addition of a scheduled non-opioid pain regimen will decrease the use and risk of opioid pain medications as well as improve pain control in head and neck surgery patients. Participants will be randomized to one of two pain regimens (opioid medication regimen vs combination regimen of opioid and non-opioid medications).

DETAILED DESCRIPTION:
Head and neck surgery patients have significant difficulty with pain control and the traditional opioid pain regimens can have increased risk in this patients population (namely, respiratory and airway compromise). Most of the literature for head and neck cancer patients focuses on pain management during chemoradiation therapy, but very few studies evaluate pain management in the post-operative setting. Patients with worse pain control and chronic opioid use do not score as well on quality of life questionnaires and have higher rates of depression and anxiety.

The few studies that did specifically evaluate post-operative pain showed success with a scheduled non-opioid management such as NSAIDs, acetaminophen, and gabapentin/pregabalin. In head and neck surgery patients, pre-operative gabapentin as compared to standard opioid pain medications was shown to have better pain control and less opioid requirements post operatively. Post-operative gabapentin has been studied and shows equivalent results, but has not been tested in a randomized controlled fashion and thus, more data is necessary. In another study evaluating scheduled acetaminophen vs as needed opioid pain medication in post-operative Cesarean section patients, there were similar results with improved pain control and less opioid use. NSAIDS are frequently avoided in post-surgical patients due to an increased risk of bleeding, but are frequently used in non-surgical patients and have shown significant benefit in pain control. Celecoxib is an NSAID that does not carry an increased bleeding risk and has been shown to be beneficial in pain control.

The pain management team in the UAB Department of Anesthesiology currently uses a combination regimen of opioid and non-opioid medication for their post-operative patients. This is the combination we plan to use in our treatment group. It consists of the standard dosing of oxycodone (an opioid) and acetaminophen, gabapentin and celecoxib (non-opioids) and is considered routine care for Anesthesiology's post-operative patients.

This study would be the first of its kind and potentially help determine a new post-operative pain management protocol for head and neck patients that is both more effective and less risky.

ELIGIBILITY:
Inclusion Criteria:

* age 18-69
* able to consent for themselves
* undergoing a "moderate" head and neck surgery at UAB, defined as procedures that generally require only 1-2 night stay in the hospital. For the purposes of this protocol, this will include patients undergoing neck dissections, glossectomy with primary closure, thyroidectomy, or parotidectomy

Exclusion Criteria:

* age < 18 or > 69
* unable to consent for themselves
* have a known opioid tolerance or are one a home opioid regimen prior to surgery
* known hepatic failure, renal failure, or sulfa allergy, as determined by standard of care labs drawn within 30 days of enrollment

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-11-10 (Actual); Primary Completion 2020-11-06 (Actual); Study Completion 2021-11-06 (Estimated)

PRIMARY OUTCOMES:
Participant pain control | 2 weeks
  Self-report via questionnaire of pain score, pain improvement, average pain, location of pain, and interference with daily activities

SECONDARY OUTCOMES:
Opioid medication use | 2 weeks
  Amount of opioid medication used, based on pill count

CONTACTS AND LOCATIONS:
Overall Officials: Erin Partington Buczek, MD, Principal Investigator — University of Alabama at Birmingham

IPD SHARING:
Plan to Share IPD: No
There is no current plan to share individual participant data for this protocol.